CLINICAL TRIAL: NCT06753955
Title: A Phase 1, Open-label Study to Evaluate the Safety, Tolerability, and Pharmacokinetics of a Single-dose of ART5803 Following IVIG Administration in Healthy Participants
Brief Title: Phase 1 Study of ART5803 Safety and PK After IVIG in Healthy Participants
Status: Active, not recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Arialys Therapeutics (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ART5803-102
Record Dates: First submitted 2024-12-23; First posted 2024-12-31 (Actual); Last update posted 2025-09-25 (Actual); Status verified 2025-09

CONDITIONS: Autoimmune Encephalitis Caused by N-Methyl D-Aspartate Receptor Antibody; Autoimmune Encephalitis Caused by N-Methyl D-Aspartate Receptor Antibody (Disorder); Autoimmune Encephalitis
Keywords: Anti-N-methyl-D-aspartate receptor (NMDAR); Encephalitis; Anti-N-methyl-D-aspartate receptor (NMDAR) Encephalitis; Intravenous immunoglobulin (IVIG)
MeSH Terms: conditions — Autoimmune Diseases of the Nervous System; Encephalitis | interventions — Immunoglobulins, Intravenous

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Cohort 1 (Other): IVIG IV infusion (not experimental) followed by ART5803 IV infusion (experimental)
  Interventions: Drug: ART5803; Drug: Intravenous immunoglobulin (IVIG)

INTERVENTIONS:
Drug: ART5803 — A monovalent (one-armed) antibody, that binds to the NTD of the NMDAR NR1 subunit without causing NMDAR inhibition, activation, or receptor internalization, while simultaneously blocking the ability of the pathogenic anti-NMDAR autoantibodies to bind to the receptor.
Drug: Intravenous immunoglobulin (IVIG) — Administered as background treatment prior to the investigational product

SUMMARY:
This study will evaluate the safety, tolerability, and pharmacokinetics (PK) of ART5803 following IVIG administration in healthy participants to investigate the potential interactions between ART5803 and IVIG

DETAILED DESCRIPTION:
Anti-N-methyl-D-aspartate receptor (NMDAR) encephalitis is one of the most common causes of autoimmune encephalitis. The disease is caused by the development of autoantibodies against the amino (N)-terminal domain (NTD) of the NMDAR subunit 1 (NR1) that bind and cross link the receptors, leading to receptor internalization and loss of function.

Arialys has developed a monovalent (one-armed) antibody, ART5803, that binds to the NTD of the NMDAR NR1 subunit without causing NMDAR inhibition, activation, or receptor internalization, while simultaneously blocking the ability of the pathogenic anti-NMDAR autoantibodies to bind to the receptor.

In treating anti-NMDAR encephalitis, intravenous immunoglobulin (IVIG) is commonly administered in conjunction with corticosteroids. Consequently, it is anticipated that IVIG may be administered to the target population prior to ART5803. IVIG has a long half-life and competitive binding of IVIG to the neonatal fragment crystallization receptor (FcRn) may result in FcRn saturation. This can potentially lead to increased clearance and/or impaired tissue distribution of ART5803 and decrease the cerebrospinal fluid (CSF) exposure to ART5803 through competition on FcRn at the blood-brain barrier (BBB).

ELIGIBILITY:
Inclusion Criteria:

1. The participant must be willing and able to provide written, signed informed consent after the nature of the study has been explained and prior to any research-related procedures.
2. The participant is a male or female, 18 to 65 years of age (inclusive) at the time of informed consent, and has a body mass index (BMI) between 18 and 32 kg/m2 (inclusive) and a weight not exceeding 100 kg.
3. The participant is healthy, as determined by medical history, physical examinations, and the clinical Investigator's judgment.
4. The participant must be willing and able to comply with all study procedures.
5. Sexually active female participants of childbearing potential and male participants with female partner(s) of childbearing potential must be willing to use a highly effective method of contraception while participating in the study. The contraceptive methods used for male and female participants must be documented in the source documents.
6. Female participants of childbearing potential must have a negative pregnancy test at Screening and be willing to have additional pregnancy tests during the study. Females considered not of childbearing potential include those who are surgically sterile (surgical bilateral oophorectomy, bilateral salpingectomy, or hysterectomy) confirmed by medical history or are post-menopausal (i.e., no menstrual bleeding for more than 12 months without an alternative medical cause and confirmation with more than 1 follicle-stimulating hormone measurement of at least > 40 IU/L [or higher per local institutional guidelines]).Women of non-childbearing potential are not required to use any contraceptive method.
7. Male participants with female partners of childbearing potential must agree to use highly effective methods of contraception, from study drug administration until at least 90 days after the last study drug administration.
8. Male participants must agree not to donate sperm, and female participants must agree not to donate eggs for the duration of the study and until at least 90 days after the last study drug administration.
9. Participants must agree not to donate blood for at least 3 months after the end-of-study (EOS) visit.

Exclusion Criteria:

1. The participant is pregnant or breastfeeding at Screening or planning to become pregnant (self or partner) at any time during the study.
2. The participant has used an investigational product or medical device within 30 days of Screening or for significant illness, such as cardiovascular, neurologic, pulmonary, hepatic, renal, metabolic, gastrointestinal, urologic, immunologic, endocrine, or psychiatric disease or disorder, or other abnormality, which may interfere with the evaluation or administration of the study drug, interpretation of participant safety or study results, or would make participation in the study an unacceptable risk including any significant acute or chronic medical condition. The Investigator is responsible for assessing the clinical significance of findings from health assessments and evaluations; however, consultation with the medical monitor may be warranted.
3. Has a concurrent disease or condition that, in the view of the Principal Investigator, places the participant at high risk of poor treatment compliance or of not completing the study, or would interfere with study participation or would affect safety. Participants with fully resolved childhood asthma with no reoccurrences or hospitalizations remain eligible for participation.
4. The participant is a regular smoker (cigarettes, e-cigarettes, and vaping included), defined as smoking daily. Participants who are non-daily smokers (up to ≤5 cigarettes per week [or vaping or e-cigarette equivalent]) are permitted to participate in the study and must agree to refrain from smoking during the in-patient stays.
5. The participant has a contraindication to undergo LP, including international normalized ratio (INR) >1.4 or other coagulopathy, platelet cell count of <120,000/µL, infection at the desired LP site, current use of anti-coagulant medication except for low dose acetylsalicylic acid, degenerative arthritis, spinal scoliosis, back surgery, suspected increased intracranial pressure on history or neurologic examination, non-communicating hydrocephalus or intracranial mass, or prior history of spinal mass or trauma.
6. The participant has a severe drug allergic history or anaphylaxis to 2 or more food products or medicines (including known sensitivity to acetaminophen/paracetamol, diphenhydramine or equivalent antihistamine, methylprednisolone or equivalent glucocorticoid, or lidocaine).
7. The participant has a known history of allergy or reaction to any component of the investigational agent formulation or IVIG or any of its components, or a history of anaphylaxis or severe systemic reaction to blood products or following any biologic therapy.
8. The participant has a history of alcohol abuse or drug addiction in the past 12 months.
9. The participant has undergone significant trauma or major surgery within 4 weeks of Screening.
10. The participant has had a vaccination with live virus, attenuated live virus, or any live viral components within 2 weeks prior to study drug administration or is planning to receive these vaccines at any time during the study and up to 8 weeks following the last study drug administration.
11. The participant has ANY of the following abnormalities in clinical laboratory tests at Screening, as assessed by the study-specific laboratory and confirmed by a single repeat if deemed necessary:

    1. Serum creatinine level more than 1.25×upper limit of normal (ULN) or an estimated glomerular filtration rate value <80 mL/min/1.73 m2 calculated with the Chronic Kidney Disease Epidemiology Collaboration formula and more than trace protein in urine.
    2. Total bilirubin, aspartate aminotransferase (AST) or alanine aminotransferase (ALT) values more than >2×ULN. Note: participants with a history of Gilbert's syndrome are excluded from participation in the study.
    3. Hematological or coagulation values outside the normal reference range for local laboratory results unless regarded as not clinically significant.
    4. Confirmed positive test for hepatitis B serology (hepatitis B surface antigen and core antibody) and/or hepatitis C polymerase chain reaction.
    5. Values indicating a deficiency of immunoglobulin A (IgA) or anti-IgA antibodies.
12. The participant has a 12-lead ECG demonstrating an abnormal corrected QT interval by Fridericia (QTcF) (>450 ms for males, >470 ms for females) or a QRS interval >120 ms. If QTcF is abnormal (>450 ms for males, >470 ms for females) or a QRS interval >120 ms, the ECG should be repeated 2 more times, and the average of the 3 QTcF or QRS interval values (i.e., the initial reading plus 2 repeats for a total of 3 readings, averaged) should be used to determine the participant's eligibility.
13. The participant has Investigator determined coronavirus disease of 2019 (COVID 19) within 4 weeks prior to Day 1, received the COVID-19 vaccine within 2 weeks prior to study drug administration, or plans to receive a COVID-19 vaccine within 9 weeks after study drug administration. Regional and site COVID-19 testing policies should be followed throughout the study.
14. The participant has a positive urine or blood result for drugs of abuse (defined as any illicit drug use) at Screening or Check-in (Day -1).
15. The participant has received any NMDAR modulator other than the study drug (e.g., ketamine, memantine, dextromethorphan, amantadine, ifenprodil, phencyclidine [PCP], acamprosate, D-cycloserine) or IVIG from within 30 days or 5 half lives of the other NMDAR modulator or IVIG (whichever is longer) of study drug administration until the end of the study.
16. The participant has a known history of primary immunodeficiency (congenital or acquired) or an underlying condition such as human immunodeficiency virus infection.
17. The participant has had a bacillus of Calmette and Guérin vaccine within 1 year of enrollment.
18. The participant has a history of severe depression, bipolar disease, or schizophrenia.
19. The participant has a risk of suicide per the C-SSRS (a score of 4 or 5 on ideation or any suicidal behavior) or, according to the Investigator's clinical judgment, has made a suicide attempt in the previous 6 months, or has a history of deliberate self-harm in the past 6 months.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 6 (Estimated)
Dates: Start 2025-03-18 (Actual); Primary Completion 2025-08-19 (Actual); Study Completion 2025-12-24 (Estimated)

PRIMARY OUTCOMES:
Safety will be assessed by the incidence and severity of treatment-emergent adverse events (TEAEs) | 13 Weeks
  ART5803 safety, as measured by the number of treatment emergent adverse events
Safety will be assessed by clinically significant changes in physical and neurological examination findings | 13 Weeks
  ART5803 safety, will be assessed by clinically significant changes in physical and neurological examination findings
Safety by assessed by clinically significant changes in vital signs | 13 Weeks
  ART5803 safety, will be assessed by clinically significant changes in vital signs including systolic and diastolic blood pressure, pulse rate, respiration rate, and body temperature
Safety by assessed by clinically significant changes in clinical laboratory outcomes | 13 Weeks
  ART5803 safety, will be assessed by clinically significant changes in clinical laboratory outcomes including clinical chemistry, hematology, coagulation, and urinalysis
Safety by assessed by clinically significant changes in 12-lead ECG findings | 13 Weeks
  ART5803 safety, will be assessed by clinically significant changes 12-lead ECG findings
Safety by assessed by clinically significant changes in concomitant medications | 13 Weeks
  ART5803 safety, will be assessed by clinically significant changes in concomitant medications
Safety by assessed by clinically significant changes in presence of anti-drug antibodies (ADAs) | 13 Weeks
  ART5803 safety, will be assessed by clinically significant changes in presence of anti-drug antibodies (ADAs)
Safety will be assessed by incidence of dose-limiting toxicity (DLTs) | 13 Weeks
  ART5803 safety, will be assessed by incidence of dose-limiting toxicity (DLTs)
Safety will be assessed by change in suicidal tendency measured by Columbia-Suicide Severity Rating Scale (C-SSRS) | 13 Weeks
  ART5803 safety, will be assessed by change in suicidal tendency as measured by the incidence of positive responses (Yes) to Item 4 or 5 on the Columbia-Suicide Severity Rating Scale (C-SSRS)
To assess the pharmacokinetics (PK) of single IV dose of ART5803 following prior doses of IVIG | 13 Weeks
  To characterize and compare the PK profile of single IV dose of ART5803 following prior doses of IVIG as measured by maximum concentration (Cmax)
To assess the pharmacokinetics (PK) of single IV dose of ART5803 following prior doses of IVIG | 13 Weeks
  To characterize and compare the PK profile of single IV dose of ART5803 following prior doses of IVIG as measured by last time point with measurable concentration (Clast)
To assess the pharmacokinetics (PK) of single IV dose of ART5803 following prior doses of IVIG | 13 Weeks
  To characterize and compare the PK profile of single IV dose of ART5803 following prior doses of IVIG as measured by minimum concentration (Cmin)
To assess the pharmacokinetics (PK) of single IV dose of ART5803 following prior doses of IVIG | 13 Weeks
  To characterize and compare the PK profile of single IV dose of ART5803 following prior doses of IVIG as measured by time at which Cmax is observed (tmax)
To assess the pharmacokinetics (PK) of single IV dose of ART5803 following prior doses of IVIG | 13 Weeks
  To characterize and compare the PK profile of single IV dose of ART5803 following prior doses of IVIG as measured by time at which Clast is observed (tlast)
To assess the pharmacokinetics (PK) of single IV dose of ART5803 following prior doses of IVIG | 13 Weeks
  To characterize and compare the PK profile of single IV dose of ART5803 following prior doses of IVIG as measured by area under the curve from time 0 to the last measurable concentration (AUC0-t)
To assess the pharmacokinetics (PK) of single IV dose of ART5803 following prior doses of IVIG | 13 Weeks
  To characterize and compare the PK profile of single IV dose of ART5803 following prior doses of IVIG as measured by area under the curve from time 0 extrapolated to infinity (AUC0-∞)
To assess the pharmacokinetics (PK) of single IV dose of ART5803 following prior doses of IVIG | 13 Weeks
  To characterize and compare the PK profile of single IV dose of ART5803 following prior doses of IVIG as measured by the half-life (t½)
To assess the pharmacokinetics (PK) of single IV dose of ART5803 following prior doses of IVIG | 13 Weeks
  To characterize and compare the PK profile of single IV dose of ART5803 following prior doses of IVIG as measured by the volume of distribution (Vd)
To assess the pharmacokinetics (PK) of single IV dose of ART5803 following prior doses of IVIG | 13 Weeks
  To characterize and compare the PK profile of single IV dose of ART5803 following prior doses of IVIG as measured by by clearance (CL)
To assess the pharmacokinetics (PK) of single IV dose of ART5803 following prior doses of IVIG | 13 Weeks
  To asses the CSF/serum ratio of ART5803 at multiple time points

SECONDARY OUTCOMES:
To assess the immunogenicity of a single IV dose of ART5803 following prior doses of IVIG | 13 Weeks
  To assess the incidence of anti-drug antibodies (ADAs) in serum from a single IV dose of ART5803 following prior doses of IVIG

OTHER OUTCOMES:
To assess changes in cognition as measured by the Mini-Mental State Examination (MMSE) after a single IV dose of ART5803 following prior doses of IVIG | 13 Weeks
  To assess the change in MMSE total scores from baseline
To assess changes in cognition as measured by the Trial Making Test Part A & B (TMT-A and TMT-B) after a single IV dose of ART5803 following prior doses of IVIG | 13 Weeks
  To assess the change in TMT-A and TMT-B total scores from baseline

CONTACTS AND LOCATIONS:
Overall Officials: Sankalp Gokhale, MD, MBA, Study Chair — Arialys Therapeutics
Locations (1):
- Nucleus Network Pty Ltd, Melbourne, Victoria, Australia

IPD SHARING:
Plan to Share IPD: No